CLINICAL TRIAL: NCT00610233
Title: Effect of Deep Brain Stimulation (DBS) on Lower Urinary Tract (LUT) Function
Brief Title: Effect of Deep Brain Stimulation on Lower Urinary Tract Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Thomas M. Kessler, MD, Department of Urology, University of Bern, 3010 Switzerland
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK 33/05; 1005
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Movement Disorder; Urinary Tract Disease
Keywords: deep brain stimulation; urodynamics
MeSH Terms: conditions — Movement Disorders; Urologic Diseases | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Urodynamic investigation with deep brain stimulation ON
  Interventions: Procedure: deep brain stimulation ON
- B (Experimental): Urodynamics with deep brain stimulation OFF
  Interventions: Procedure: Deep brain stimulation OFF

INTERVENTIONS:
Procedure: deep brain stimulation ON — deep brain stimulation in the ON state
  Arms: A
Procedure: Deep brain stimulation OFF — Urodynamic investigation with deep brain stimulation in the OFF state
  Arms: B

SUMMARY:
The precise mechanisms underlying cerebral regulation of lower urinary tract (LUT) function are still poorly understood. Patients with deep brain stimulation (DBS) offer the unique opportunity to investigate the role of different cerebral centers on LUT function.

We hypothesize that DBS has a significant effect on LUT function and that these effects depend on the specific stimulated cerebral center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with deep brain stimulation (DBS)

Exclusion Criteria:

* Pregnancy
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Effect of deep brain stimulation (DBS) on urodynamic parameters | immediately and 3 months after study inclusion

SECONDARY OUTCOMES:
Changes in questionnaire data due to deep brain stimulation (DBS) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Kessler, MD, Principal Investigator — Department of Urology, University of Bern, 3010 Switzerland
Locations (2):
- Switzerland (2):
  - Department of Neurology, University of Bern, Bern
  - Department of Urology, University of Bern, Bern